CLINICAL TRIAL: NCT05714306
Title: Phase I/II Study to Test the Immunogenicity, Feasibility, and Safety of Autologous PEP-DC Vaccine vs. Autologous OC-DC Vaccine Followed by PEP-DC Vaccine, in Combination With Low-dose Cyclophosphamide, in Patients With Advanced HGSOC
Brief Title: PEP-DC and OC-DC Vaccine in High Grade Serous Ovarian Carcinoma
Acronym: CHUV-OVACURE
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Lack of funding
Sponsor: Centre Hospitalier Universitaire Vaudois (Other)
Responsible Party: Principal Investigator, Dr. Apostolos Sarivalasis, MD, Associate Physician, Centre Hospitalier Universitaire Vaudois
Allocation: Not Applicable | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CHUV-DO-0005-OVACURE_2017
Record Dates: First submitted 2023-01-17; First posted 2023-02-06 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-03

CONDITIONS: Ovarian Carcinoma
Keywords: advanced high grade serous ovarian carcinoma; dendritic cell vaccine
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A - PEP-DC1 + low dose cyclophosphamide (Experimental): In arm A, patients will receive PEP-DC1 vaccine in combination with low dose cyclophosphamide.
  Interventions: Biological: PEP-DC1; Drug: Low dose cyclophosphamide
- Arm B - OC-DC + low dose cyclophosphamide followed by PEP-DC2 + low dose cyclophosphamide (Experimental): In arm B, patients will receive first, the OC-DC vaccine in combination with low dose cyclophosphamide, then PEP-DC2 vaccine in combination with low dose cyclophosphamide. Finally, patients will be vaccinated with the personalized PEP-DC2 to continue maintenance vaccination.
  Interventions: Biological: OC-DC; Biological: PEP-DC2; Drug: Low dose cyclophosphamide

INTERVENTIONS:
Biological: PEP-DC1 — PEP-DC1 vaccine comprises autologous dendritic cells pulsed with personalized peptides detected or predicted a priori (using our current integrated antigen identification methodologies).
  Arms: Arm A - PEP-DC1 + low dose cyclophosphamide
Biological: OC-DC — OC-DC vaccine is an autologous dendritic cell vaccine loaded with autologous oxidized tumor lysate.
  Arms: Arm B - OC-DC + low dose cyclophosphamide followed by PEP-DC2 + low dose cyclophosphamide
Biological: PEP-DC2 — PEP-DC2 comprises autologous dendritic cells pulsed with the peptides detected or predicted after vaccination with OC-DC.
  Arms: Arm B - OC-DC + low dose cyclophosphamide followed by PEP-DC2 + low dose cyclophosphamide
Drug: Low dose cyclophosphamide — Cyclophosphamide administered on D1 of each cycle, the day prior to each vaccination (Vx) at a dose of 200 mg/m2 intravenously (i.v.)

SUMMARY:
Single center, phase I/II randomized 2-arm study, evaluating two different vaccination regimens combined with low-dose cyclophosphamide in patients with advanced high grade serous ovarian carcinoma (HGSOC):

* Arm A patients will be vaccinated with a personalized peptide vaccine comprised of autologous monocyte-derived dendritic cells (moDC) loaded with patient-specific peptides (PEP-DC1 vaccine) identified a priori at screening (8 patients);
* Arm B patients will be vaccinated with a personalized tumor lysate vaccine comprising autologous moDC loaded with patient-specific autologous oxidized tumor lysate (OC-DC vaccine), followed by PEP-DC2 vaccine comprised of autologous moDC loaded with up to 10 patient-specific peptides identified midway through OC-DC vaccination (8 patients).

In both arms, patients will receive a low dose cyclophosphamide the day before vaccination. Patients will be vaccinated after the end of adjuvant platinum-based chemotherapy, until vaccine exhaustion, disease recurrence, major toxicity or patient withdrawal, whichever is earlier.

DETAILED DESCRIPTION:
This will be a single center, Phase I/II randomized, two-arm, open-label study to evaluate immunogenicity, safety, and feasibility of two different vaccination regimens combined with low-dose cyclophosphamide in patients with surgically resected, advanced HGSOC. Patients with HGSOC at International Federation of Gynecology and Obstetrics (FIGO) stage III or IV who completed either primary debulking surgery (PDS) or interval debulking surgery (IDS) without residual disease (R0) and who have received at least 6 cycles of adjuvant standard of care (SOC) platinum-based chemotherapy after PDS, or 3 cycles of platinum-based perioperative chemotherapy within an IDS will be eligible for this protocol. A total of 16 patients (8 patients in each arm) will be randomized 1:1 as follows:

* In arm A, patients will receive PEP-DC1 vaccine comprising autologous dendritic cells pulsed with personalized peptides detected or predicted a priori (using our current integrated antigen identification methodologies).
* In arm B, patients will receive first, the OC-DC vaccine, an autologous dendritic cell vaccine loaded with autologous oxidized tumor lysate. Then, tumor antigens specifically recognized by the patients' immune response induced by OC-DC vaccination will be identified/predicted using integrated methodologies to enable production of PEP-DC2 vaccine (autologous dendritic cells pulsed with the peptides detected or predicted after vaccination with OC-DC). Finally, patients will be vaccinated with the personalized PEP-DC2 to continue maintenance vaccination.

In both arms, vaccines will be administered to the patients in combination with low dose cyclophosphamide the day before vaccination. Patients will be vaccinated in the adjuvant setting, with first vaccine injected no more than 18 weeks after the end of SOC platinum-based chemotherapy. Patients will be vaccinated until vaccine exhaustion (which may happen any time after dose 6), disease recurrence, major toxicity or patient withdrawal, whichever is earlier.

ELIGIBILITY:
Patient enrollment will follow a two-step procedure (at screening before randomization and at assessment after vaccine production) of conditions required for initiating vaccination. Patients must meet all of the criteria described in this section prior to receiving any vaccination.

AT SCREENING:

Inclusion Criteria:

1. Signed Informed Consent Form
2. Histologically confirmed diagnosis of advanced, FIGO stage III or IV, high grade serous ovarian carcinoma (HGSOC)
3. Underwent PDS or IDS without macroscopic residual disease, (R0)
4. a. Received at least 3 cycles of peri-operative platinum-based chemotherapy before IDS, with the intention to complete at least 6 cycles of peri-operative platinum-based chemotherapy.

   OR b. Has completed 6 cycles of adjuvant platinum-based chemotherapy after PDS. In case of toxicity prohibiting 6 cycles of adjuvant platinum-based chemotherapy, a minimum of 4 cycles are required.
5. Tumor material is available and sufficient for both OC-DC preparation and identification of Top 10 personalized peptides (PEPs) required for PEP-DC vaccine preparation.
6. Age ≥18 years.
7. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
8. Willing and able to comply with study procedures
9. Has adequate hematologic and end organ function (kidney, liver and bone marrow), defined by the following laboratory results (complete blood count (CBC), enzyme tests) obtained within 14 days prior to randomization:

   * Hemoglobin ≥ 80 g/L
   * Neutrophil count ≥ 1.0 x G/L (independently of administration of growth factor within 4 weeks prior to randomisation)
   * Platelet count ≥ 100 G/L
   * Serum creatinine ≤ 1.5x Institutional Upper Limit of Normal (ULN) or Creatinine Clearance ≥ 40 mL/min.
   * Serum bilirubin ≤ 1 ULN (except subjects with Gilbert's syndrome who must have a total bilirubin level of <3.0 x ULN)
   * aspartate aminotransferase (AST) / alanine transaminase (ALT) ≤ 3 x ULN
   * Alkaline phosphatase ≤ 1.5 x ULN
   * Coagulation: International Normalized Ratio (INR) or Prothrombin Time (PT) ≤ 1.5 X ULN unless subject is receiving anticoagulant therapy as long as PT or partial thromboplastin time (PTT) is within therapeutic range of intended use of anticoagulants; activated Partial Thromboplastin Time (aPTT) ≤ 1.5 X ULN unless subject is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants.
10. Has adequate serology defined by the following laboratory results obtained within 14 days prior to randomization:

    * Negative test for Human Immunodeficiency Virus (HIV)
    * Patients with active or chronic hepatitis B (defined as having a positive hepatitis B surface antigen [HBsAg] test at screening) are not eligible.

      * Patients with past/resolved Hepatitis B Virus (HBV) infection (defined as having a negative HBsAg test and a positive antibody to hepatitis B core antigen (anti-HBc) antibody test) are eligible, if HBV Deoxyribonucleic Acid (DNA) test is negative.
      * HBV DNA must be obtained in patients with positive hepatitis B core antibody prior to start of study treatment.
    * Patients with active hepatitis C are not eligible. Patients positive for Hepatitis C Virus (HCV) antibody are eligible only if Polymerase Chain Reaction (PCR) is negative for HCV Ribonucleic Acid (RNA).
11. Absence of any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol.
12. Patient is able to undergo leukapheresis

Exclusion Criteria:

1. A secondary debulking surgery is foreseen.
2. Prior exposure to anti-Cytotoxic T-Lymphocyte-Associated Protein 4 (CTLA4) and anti-Programmed cell Death 1 (PD1) / anti-Programmed cell Death Ligand (PD-L1) antibodies or other immunotherapy.
3. Woman of child-bearing potential (WOCBP). By definition, all patients with HGSOC of FIGO stage III to IV who have undergone PDS or IDS, will have undergone total hysterectomy with bilateral salpingo-oophorectomy, and will therefore be women without child-bearing potential. Therefore, no pregnancy tests have to be performed because no WOCBP will be enrolled in this trial.
4. Breastfeeding women
5. Other malignancy within 2 years prior to randomization, except for those (for example ductal carcinoma in situ of breast and cervical intraepithelial neoplasia) treated with curative intent. Patients with a predicted 5-year recurrence-free survival rate ≥95% can be included at the investigator's discretion.
6. Patients with diagnosis of paraneoplastic syndrome.
7. Current, recent (within 4 weeks prior to randomization), or planned participation in an experimental drug study.
8. Patient has a serious, non-healing wound, ulcer, or bone fracture.
9. Patients with Glucose-6-phosphate dehydrogenase (G6PD) deficiency are excluded. Patients with high bleeding risk or any other hereditary coagulation disorder can be enrolled after careful evaluation, at principal investigator (PI)'s discretion.
10. Past history with cardiac or vascular problems:

    1. New York Heart Association Class II or greater congestive heart failure
    2. History of myocardial infarction or unstable angina within 6 months prior to randomization
    3. History of stroke or transient ischemic attack within 6 months prior to randomization
    4. Significant vascular disease (e.g., aortic aneurysm requiring surgical repair or recent peripheral arterial thrombosis) within 6 months prior to randomization
    5. Evidence of bleeding diathesis or significant coagulopathy (in the absence of therapeutic anticoagulation)
    6. Patient has a grade II or greater peripheral vascular disease.
    7. Patient has a clinically significant peripheral artery disease, e.g., those with claudication, within 6 months prior to randomisation.
11. Any other diseases, metabolic dysfunction, physical examination findings, or clinical laboratory findings giving reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug or that may affect the interpretation of the results or render the patient at high risk from treatment complications.
12. Patient has organ allografts.
13. Known hypersensitivity to any component of the study treatment
14. History of autoimmune disease, including but not limited to myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, vascular thrombosis associated with antiphospholipid syndrome, Wegener's granulomatosis, Sjögren's syndrome, Guillain-Barré syndrome, multiple sclerosis, vasculitis, or glomerulonephritis.

    1. Patients with a history of autoimmune-related hypothyroidism on a stable dose of thyroid replacement hormone are eligible for this study.
    2. Patients with controlled Type I diabetes mellitus on a stable insulin regimen are eligible
15. Administration of a live, attenuated vaccine within 8 weeks before randomization. Exception: Influenza vaccination should be given during influenza season only (approximately October to March). Patients must not receive live, attenuated influenza vaccine within 4 weeks prior to randomization.
16. History of immediate hypersensitivity reaction to streptomycin and penicillin.

AT VACCINATION:

Inclusion Criteria:

1. Has received 6 cycles of platinum-based chemotherapy to first vaccination (minimum of 4 cycles platinum-based chemotherapy in case of severe toxicity and inability to administer all planned 6 cycles).
2. Confirmation from the Centre des Thérapies Experimentales (CTE) cellular manufacturing facility that at least 6 doses of vaccines have been produced for the patient (for Arm A: PEP-DC1 vaccines, Arm B: OC-DC vaccines) at the CTE cellular manufacturing facility.

   Has adequate hematologic and end organ function (kidney, liver and bone marrow), defined by the following laboratory results (complete blood count [CBC], enzyme tests) obtained before start of the study treatment:
   * Hemoglobin ≥ 80 g/L
   * Neutrophil count ≥ 1.5 x G/L
   * Platelet count ≥ 100 G/L
   * Serum creatinine, ≤ 1.5x Institutional Upper Limit of Normal (ULN) or Creatinine Clearance ≥ 40 mL/min, calculated using the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) formula
   * Serum bilirubin ≤ 1 ULN (except subjects with Gilbert's syndrome who must have a total bilirubin level of <3.0 x ULN )
   * AST/ALT ≤ 3 x ULN
   * Alkaline phosphatase ≤ 1.5 x ULN
   * Coagulation: International Normalized Ratio (INR) or Prothrombin Time (PT) ≤ 1.5 X ULN unless subject is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants; Activated Partial Thromboplastin Time (aPTT) ≤ 1.5 X ULN unless subject is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants.
3. Has no evidence of disease confirmed by computerized tomography (CT)-scan of chest/abdomen/pelvis (i.e. tumor-free by CT scan according to RECIST v1.1) and CA 125 Gynecologic Cancer InterGroup (GCIC) criteria (i.e. normal CA 125 blood level) before start of the study treatment.
4. Has recovered from any toxic effects of prior chemotherapy to ≤ Grade 1 per the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE v.5.0) except for toxicities described below, as long as they do not put at risk the patient's condition and do not require systemic immunosuppressive steroids at any dose, including but not limited to:

   * Fatigue
   * Alopecia
   * Skin disorders
   * Stable neuropathy
   * Endocrinopathies requiring replacement treatment Note: For other medical conditions, or for any other toxicity with a higher grade but controlled by adequate treatment, prior discussion and agreement with the sponsor is mandatory.

Exclusion Criteria:

1. Treatment with systemic immunosuppressive medications (including but not limited to prednisone, dexamethasone, cyclophosphamide, azathioprine, methotrexate, thalidomide, and anti-tumor necrosis factor (anti-TNF) agents) within 4 weeks prior to first study treatment.

   Exceptions:
   * Patients who are receiving acute, low-dose, systemic immunosuppressant medications (e.g., a one-time dose of dexamethasone for nausea) or physiologic replacement doses (i.e., prednisone 5-7.5 mg/day, or other) for adrenal insufficiency may be enrolled in the study.
   * The use of inhaled corticosteroids and mineralocorticoids (e.g., fludrocortisone) is allowed.
   * Standard premedication of paclitaxel, docetaxel, nab-paclitaxel, or Caelyx (pegylated liposomal doxorubicin i.e. PLD).

     1. When tri-weekly 175 mg/m2 paclitaxel is given: 20mg of dexamethasone administered 12 hours and 6 hours before paclitaxel administration (or according to Institution's guidelines) during last chemotherapy cycle (C6D1) is allowed.
     2. When weekly 80 mg/m2 paclitaxel is given: on the day of treatment, administration of a single 8 mg dose of dexamethasone before paclitaxel administration is allowed.
   * Treatment of late onset nausea and treatment of allergic reaction induced by SOC chemotherapy
2. Administration of a live, attenuated vaccine within 8 weeks before start of study treatment. Exception: Influenza vaccination should be given during influenza season only (approximately October to March). Patients must not receive live, attenuated influenza vaccine within 4 weeks prior to start of study treatment.
3. Any other diseases, cardiac, metabolic or other dysfunction, physical examination findings or clinical laboratory findings since the screening visit giving reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug or that may affect the interpretation of the results or render the patient at high risk from treatment complications.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-08-01 (Estimated); Primary Completion 2030-03 (Estimated); Study Completion 2030-03 (Estimated)

PRIMARY OUTCOMES:
Immunogenicity of OC-DC + PEP-DC vaccine vs. PEP-DC vaccine | through study completion, an average of 7 years
  The number of personalized tumor antigen (PTAs) ranked as Top 100 will be identified for each patient before and after treatment and the difference will be compared between the two arms at least at two time-points, first at the end of the 3rd cycle (C3W3), and second, at end of treatment (EOT) visit (if possible at C6W4-W6 also). Specifically, an immunogenicity scoring will be determined as follows: for each of the 100 pre-determined top PTAs, a score will indicate how many peptides either become newly detected (shift from undetectable to detectable) or have a magnitude (frequency of T-cell directed against the epitope) increased by ≥ 2 fold.

SECONDARY OUTCOMES:
Feasibility of vaccines production and administration in each arm | 3 years after study activation
  Feasibility of producing and administering vaccines will be evaluated by:
  i) the number of patients for whom vaccine is produced successfully (defined as production and quality control release of at least 6 doses of PEP-DC1 vaccine for Arm A patients, and at least 6 doses of OC-DC vaccine and 6 doses of PEP-DC2 vaccine for Arm B patients) and ii) the number of patients who receive at least one vaccine dose among the randomized patients.
  Feasibility is considered as achieved if within each arm, at least 50% of the randomized subjects comply with these criteria.
Assessment of adverse events in each treatment arm | From signature of informed consent form (ICF) until 30 days after the last treatment (vaccine/cyclophosphamide)
  Collection of adverse events and serious adverse events, and treatment limiting toxicities
Time to progression (TTP) | 5 years
  Will be evaluated in the 2 arms. TTP is the time from randomization to date of first documented objective tumor progression according to RECIST 1.1 criteria and cancer antigen (CA) 125 Gynecologic Cancer InterGroup (GCIG) criteria.
Disease free survival (DFS) rate | Evaluated at 12, 24, and 36 months
  DFS is defined as the time from randomization to date of first documented objective tumor recurrence according to RECIST 1.1 and CA 125 GCIG criteria, or, death due to any cause or last patient contact in which the patient was determined to be disease-free.
Overall survival (OS) | Evaluated at 5 years
  Will be assessed in both arms. OS is defined as the time from randomization to date of death due to any cause, or last patient contact.

CONTACTS AND LOCATIONS:
Overall Officials: Apostolos Sarivalasis, MD, Principal Investigator — Centre Hospitalier Universitaire Vaudois; Lana Kandalaft, Pharm D, PhD, Study Chair — Centre Hospitalier Universitaire Vaudois